CLINICAL TRIAL: NCT00425906
Title: A Pilot Study of Nicotine for "Hunger Pain" in Patients With Bowel Obstruction From Incurable Cancer
Brief Title: Nicotine in Treating "Hunger Pain" in Patients With Malignant Bowel Obstruction Caused By Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patient enrollment occurred.
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Aminah Jatoi, M.D., Mayo Clinic
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000526182; P30CA015083 (NIH); MC03C2 (Other: Mayo Clinic Cancer Center); 1217-03 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2007-01-19; First posted 2007-01-23 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2011-07

CONDITIONS: Anorexia; Constipation, Impaction, and Bowel Obstruction; Pain; Psychosocial Effects of Cancer and Its Treatment; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: psychosocial effects of cancer and its treatment; unspecified adult solid tumor, protocol specific; constipation, impaction, and bowel obstruction; anorexia; pain
MeSH Terms: conditions — Anorexia; Constipation; Intestinal Obstruction; Pain | interventions — Nicotine; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicotine inhaler (Experimental)
  Interventions: Drug: nicotine; Procedure: Quality of life
- Placebo inhaler (Placebo Comparator)
  Interventions: Other: Placebo; Procedure: Quality of life

INTERVENTIONS:
Drug: nicotine
  Arms: Nicotine inhaler
Other: Placebo
  Arms: Placebo inhaler
Procedure: Quality of life

SUMMARY:
RATIONALE: The use of a nicotine inhaler may help decrease appetite and relieve "hunger pain" (an intense craving for food) in patients with malignant bowel obstruction caused by cancer.

PURPOSE: This randomized clinical trial is studying the side effects and how well a nicotine inhaler works in treating "hunger pain" in patients with malignant bowel obstruction caused by cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether patients with malignant bowel obstruction due to incurable cancer utilize a potential therapy for "hunger pain."
* Determine, preliminarily, the efficacy and toxicity of nicotine in treating "hunger pain" in these patients.
* Determine whether nicotine results in a decline in circulating ghrelin (for patients enrolled at the Mayo Rochester Clinic only).
* Evaluate hormonal changes in patients treated with nicotine (for patients enrolled at the Mayo Rochester Clinic only).

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter, pilot study. Patients are stratified according to vomiting status within the past 24 hours (yes vs no) and use of narcotics (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive a nicotine inhaler to use as needed for "hunger pain." Treatment continues for up to 48 hours in the absence of unacceptable toxicity .
* Arm II: Patients receive a placebo inhaler to use as needed for "hunger pain." Treatment continues for up to 48 hours in the absence of unacceptable toxicity.

After 48 hours, patients in arm I may continue nicotine therapy off study. Patients in arm II who are not surgical candidates may cross over to treatment with the nicotine inhaler off study.

Blood and spot urine samples are collected at baseline and after 48 hours from patients enrolled at the Mayo Rochester Clinic. Blood samples are analyzed to evaluate circulating hormone (e.g., ghrelin, leptin) concentrations. Urine samples are analyzed to evaluate nicotine and nicotine metabolite concentrations.

Global quality of life is assessed at baseline and after 48 hours. "Hunger pain" is assessed at baseline.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of any incurable malignancy
* Presence of malignant bowel obstruction
* Must be on strict "nothing per os" (NPO) status over the next 48 hours

  * Ice chips allowed
* Acknowledges that "hunger pain" is a problem

PATIENT CHARACTERISTICS:

* Mentally competent
* No history of life-threatening arrhythmia
* No severe or worsening angina
* No accelerated hypertension
* No known hypersensitivity to nicotine
* Not pregnant or nursing
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

* Concurrent short-term use of dexamethasone or other hormonal therapy or symptom control strategy allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-12

PRIMARY OUTCOMES:
Determination of whether ≥ 50% of patients utilize nicotine for treating "hunger pain" ≥ 2 times over a 48-hour period | 48 Hours

SECONDARY OUTCOMES:
Toxicity as measured by CTCAE v 2.0 | 48 hours
Global quality of life | 48 hours
Hunger assessment | 48 hours
Change in circulating hormonal concentrations (for patients enrolled at the Mayo Rochester Clinic only) | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic; Gerardo Colon-Otero, MD, Principal Investigator — Mayo Clinic